CLINICAL TRIAL: NCT03659006
Title: Identification of Predictive Neuroinflammatory Biomarkers of Neuro-radiological Evolution in Severe Traumatic Brain Injury
Acronym: ICON-TBI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Hopital Universitaire Robert-Debre (Other); University of Cambridge (Other); Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: K171201J
Record Dates: First submitted 2018-07-09; First posted 2018-09-06 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-07

CONDITIONS: Severe Traumatic Brain Injury
Keywords: inflammatory Biomarkers, Traumatic brain injury, multimodal MRI, tertiary lesion
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biological Collection (Experimental): Blood sampling on catheter and CSF sampling from VDE, multimodal MRI at D42 and D365, Neurological and neuropsychological evaluation at one year
  Interventions: Biological: Biological Collection

INTERVENTIONS:
Biological: Biological Collection — Blood sampling on catheter and CSF sampling from VDE, multimodal MRI at D42 and D365, Neurological and neuropsychological evaluation at one year

SUMMARY:
Tertiary lesions responsible of the neurological decline after severe traumatic brain injury (TBI) are partially due to a persistent neuro-inflammation directly modulated by inflammatory mediators during the acute phase and detectable by using both multimodal MRI imaging and biological biomarkers during the acute phase after traumatic brain injury.

The main objective is to identify if the level of IL-1beta in cerebrospinal fluid predict in a reliable and reproducible way, the neuro-radiological evolution evaluated by the comparison of a quantitative MRI performed in post-resuscitation and at one year (quantitative ΔIRM) in traumatic brain injuried patients.

The secondary objectives are:

* To understand the links between the acute and chronic neuro-inflammatory phase in a population of TBI,
* To explore the contribution of the adaptive immune response in the persistent activation of the immune response,
* To Examine the links between persistent neuroinflammation, clinical deterioration and neuroimaging,
* To establish a correlation between the pathology and the physio-pathology of TBI.

ELIGIBILITY:
Inclusion Criteria:

1. patient ≥ 18 years old at the time of inclusion
2. Written and informed consent obtained from the family / proxy
3. Patient hospitalized in neuro-ICU following severe TBI with GCS ≤ 8 at admission
4. Intubated / ventilated patient scheduled for external ventricular bypass within 24 hours of hospitalization
5. Absence of contraindications to perform an MRI
6. Patient affiliated to a social security scheme (free State medical aid excluded)

Exclusion Criteria:

1. Patient under protection of the law (guardianship or tutorship)
2. TBI of ballistic origin
3. Pregnant woman
4. Pre-existing cerebral disease that can bias the MRI scan evaluation
5. Contraindications to the MRI (pace maker, medical device incompatible with MRI, metal plates, ...)
6. Patient with severe impairment of vital and / or life-threatening function with disability prior TBI
7. Neurological antecedent susceptible to interfere with clinical evolution at one year
8. Severe cardiogenic shock
9. Severe respiratory impairment
10. Extra-brain injuries involving immediate life-threatening
11. Hemoglobin level below 9g / dL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-10-15 (Actual); Primary Completion 2020-07-30 (Estimated); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
Interleukin-1 level in blood predict changes in brain volume assessed by quantitative MRI. | Day 42 and 12 months
  Brain volume evolution assessed by quantitative MRI between Day 42 and Day 365

SECONDARY OUTCOMES:
Concentrations of biomarkers such as Tau protein and beta-amyloid plaques in serum and cerebrospinal fluid (Aβ1-42, T-tau, and P-tau181P and Interleukin 1) | Blood and CSF samples collected at Day1, Day2, Day3, Day5 and Day7
  Plasma and Serum biological collection, multimodal MRI database, clinical database

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Degos, PU-PH, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Anesthesy department - Hôpital Pitié Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: No